CLINICAL TRIAL: NCT04076215
Title: Measuring the Biochemical and Physiological Response to Controlled Stressogenic Stimuli
Brief Title: Biochemical and Physiological Response to Stressogenic Stimuli
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nadav Goldental (Other)
Responsible Party: Sponsor-Investigator, Nadav Goldental, Principal investigator, The Chaim Sheba Medical Center
Organization: The Chaim Sheba Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6263-19-SMC
Record Dates: First submitted 2019-08-22; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pariticapnts with PTSD (Experimental)
  Interventions: Behavioral: Stressogenic stimulus; Device: Biobeat smart watch and adhesive biosensor patches.
- Pariticapnts without PTSD (controls) (Experimental)
  Interventions: Behavioral: Stressogenic stimulus; Device: Biobeat smart watch and adhesive biosensor patches.

INTERVENTIONS:
Behavioral: Stressogenic stimulus — Participants will be exposed to an anxiety-provoking stimulus for 15-20 minutes, in a controlled setting
Device: Biobeat smart watch and adhesive biosensor patches. — Physiological and biochemical measures will be obtained using the Biobeat smart watch and adhesive biosensor patches.

SUMMARY:
Post-traumatic stress disorder (PTSD) is characterized by physiological changes, some of which are thought to be chronic, while others are observed in response to stressogenic stimuli. A psychiatric diagnosis of PTSD is currently based mainly on non-quantitative elements, such as interviews and subjective impressions. Discernable patterns of stress-related measures may constitute a physiological and biochemical phenotype characteristic of PTSD, which may serve as a biomarker and support diagnostic decisions, as well as personalized treatment plans.

The current study is aimed at examining the possibility of basing a psychiatric diagnosis by measuring changes in the biochemical phenotype of participants with PTSD. Physiological and biochemical data will be collected from participants with and without PTSD using wearable sensors and adhesive biosensor patches. The data will be collected in two conditions: in a neutral, quiet situation, and during and following exposure to controlled stressogenic stimuli.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis (excluding controls)
* Proper ability to give informed consent

Exclusion Criteria:

* Active oncological/cardiovascular condition
* Dialysis patients
* Active psychotic or suicidal symptoms
* Severe dissociative symptoms
* A traumatic brain injury (TBI) diagnosis
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Significant differences between groups - HRV | 3 hours
  Significant differences in Heart Rate Variability - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups - temperature | 3 hours
  Significant differences in physiological changes - body temperature- between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups - SPO2 | 3 hours
  Significant differences in physiological changes - Saturation SPO2- between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups - blood pressure | 3 hours
  Significant differences in physiological changes - continuous blood pressure- between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups - pulse pressure | 3 hours
  Significant differences in physiological changes - pulse pressure - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups -respiratory rate | 3 hours
  Significant differences in physiological changes - respiratory rate- between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups -stroke volume | 3 hours
  Significant differences in physiological changes - stroke volume- between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups -cardiac output | 3 hours
  Significant differences in physiological changes - cardiac output - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in physiological changes between groups - systemic vascular resistance | 3 hours
  Significant differences in physiological changes - systemic vascular resistance- between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in cortisol levels between groups | 3 hours
  Significant differences in biochemical changes - cortisol - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - C-reactive protein | 3 hours
  Significant differences in biochemical changes - C-reactive protein - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - Interleukin 6 | 3 hours
  Significant differences in biochemical changes - Interleukin 6 - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - N-terminal B-type natriuretic peptide | 3 hours
  Significant differences in biochemical changes - N-terminal B-type natriuretic peptide - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - 8-oxo-7 | 3 hours
  Significant differences in biochemical changes - 8-oxo-7- between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - 8-dihydro-2'-deoxyguanosine | 3 hours
  Significant differences in biochemical changes - 8-dihydro-2'-deoxyguanosine - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - hexanone | 3 hours
  Significant differences in biochemical changes - hexanone - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - acetic acid | 3 hours
  Significant differences in biochemical changes - acetic acid - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - heptane | 3 hours
  Significant differences in biochemical changes - heptane - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - hexanal | 3 hours
  Significant differences in biochemical changes -hexanal - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - 3-heptanone | 3 hours
  Significant differences in biochemical changes - 3-heptanone - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - hexanoic acid | 3 hours
  Significant differences in biochemical changes - hexanoic acid - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - heptanal | 3 hours
  Significant differences in biochemical changes -heptanal - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - nonanal | 3 hours
  Significant differences in biochemical changes - nonanal - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli
Significant differences in biochemical changes between groups - glucose | 3 hours
  Significant differences in biochemical changes - glucose - between groups (participants with PTSD and controls) before and after exposure to stressogenic stimuli